CLINICAL TRIAL: NCT02246764
Title: A Double-masked, Randomized, Multi-center, Active-controlled, Parallel, 12-month Study Assessing the Safety of AR-13324 Ophthalmic Solution, 0.02% QD & BID Compared to Timolol Maleate Ophthalmic Solution, 0.5% BID in Patients With Elevated Intraocular Pressure
Brief Title: Study of Netarsudil (AR-13324) Ophthalmic Solution in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS303
Record Dates: First submitted 2014-09-16; First posted 2014-09-23 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-01

CONDITIONS: Ocular Hypertension; Glaucoma
Keywords: Ocular hypertension.; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — netarsudil; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AR-13324 Ophthalmic Solution 0.02% & placebo (Experimental): 1 drop AR-13324 in the evening (PM) and 1 drop placebo in the morning (AM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%; Other: Placebo
- AR-13324 Ophthalmic Solution 0.02% BID (Experimental): 1 drop AR-13324 twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02% BID
- Timolol maleate Ophthalmic Solution 0.5% BID (Active Comparator): 1 drop Timolol maleate twice daily (BID) in the morning (AM) and evening (PM) in both eyes (OU)
  Interventions: Drug: Timolol maleate Ophthalmic Solution 0.5% BID

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.02% — 1 drop once daily (QD), PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo
Drug: AR-13324 Ophthalmic Solution 0.02% BID — 1 drop BID, AM/PM, OU
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02% BID
Drug: Timolol maleate Ophthalmic Solution 0.5% BID — 1 drop BID, AM/PM, OU
  Arms: Timolol maleate Ophthalmic Solution 0.5% BID
Other: Placebo — 1 drop QD, AM, OU
  Arms: AR-13324 Ophthalmic Solution 0.02% & placebo

SUMMARY:
The purpose of this study is to evaluate the ocular and systemic safety of Netarsudil (AR-13324) Ophthalmic Solution, 0.02% q.d. and b.i.d. for 12 months compared to the active comparator Timolol Maleate Ophthalmic Solution, 0.5%.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) IOP (Intraocular Pressure) >20 mm Hg and < 27 mm Hg in the study eye at 2 qualification visits (08:00 hr), 2-7 days apart. At second qualification visit, IOP > 17 mm Hg and < 27 mm Hg at 10:00 and 16:00 hrs (in the same eye).
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS (Early Treatment Diabetic Retinopathy Study) in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic:

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. Intraocular pressure ≥27 mm Hg (unmedicated) in both eyes (individuals who are excluded for this criterion are not allowed to attempt requalification), or use of more than two ocular hypotensive medications within 30 days of screening. Note: fixed dose combinations count as two medications.
3. Known hypersensitivity to any component of the formulations to be used (benzalkonium chloride, etc.), to topical anesthetics or β-adrenoceptor antagonists.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in either eye.
5. Refractive surgery in either eye (e.g., radial keratotomy, PRK (photorefractive keratectomy), LASIK (laser eye surgery), corneal cross-linking, etc.).
6. Ocular trauma in either eye within the six months prior to screening, or ocular surgery or non-refractive laser treatment within the three months prior to screening.
7. Recent or current evidence of ocular infection or inflammation in either eye. Current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex or zoster keratitis at screening in either eye.
8. Ocular medication in either eye of any kind within 30 days of screening, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after screening) or c) lubricating drops for dry eye (which may be used throughout the study).
9. Clinically significant ocular disease in either eye (e.g., corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (e.g., cup-disc ratio > 0.8, severe visual field defect).
10. Central corneal thickness in either eye greater than 600 µm at screening.
11. Any abnormality in either eye preventing reliable applanation tonometry of either eye.

    Systemic:
12. Clinically relevant abnormalities (as determined by the investigator) in laboratory tests at screening which may impact the study.
13. Known hypersensitivity or contraindication to beta-adrenoceptor antagonists (e.g., chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure or heart rate; second or third degree heart block or congestive heart failure; severe diabetes).
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Participation in any investigational study within 30 days prior to screening.
16. Changes of systemic medication that could have an effect on IOP within 30 days prior to screening, or anticipated during the study.
17. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals
Locations (1):
- Nancy Ramirez, Bedminster, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AR-13324 Ophthalmic Solution 0.02% & Placebo: 1 drop AR-13324 in the evening (PM) & 1 drop placebo in the morning (AM) in both eyes (OU)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | AR-13324 Ophthalmic Solution 0.02% BID | Timolol Maleate Ophthalmic Solution 0.5% BID
Started | 34 | 36 | 23
Completed | 16 | 4 | 19
Not Completed | 18 | 32 | 4
Not completed — Adverse Event | 15 | 29 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Disallowed Concomitant Medication | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Protocol Violation | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | AR-13324 Ophthalmic Solution 0.02% BID | Timolol Maleate Ophthalmic Solution 0.5% BID | Total
Number analyzed (Participants) | 34 | 36 | 23 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.73) | 64.4 (7.84) | 61.9 (12.52) | 63.8 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 8 | 44
  Male | 16 | 18 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 33 | 35 | 23 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 30 | 34 | 19 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 36 | 23 | 93

OUTCOME MEASURES:

1. Primary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups
Time Frame: 12 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: days
Groups:
- AR-13324 Ophthalmic Solution 0.02% BID: 1 drop AR-13324 twice daily (BID) in the morning and evening (PM) in both eyes (OU)
- Timolol Maleate Ophthalmic Solution 0.5% BID: 1 drop Timolol maleate twice daily (BID) in the morning and evening (PM) in both eyes (OU)
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | AR-13324 Ophthalmic Solution 0.02% BID | Timolol Maleate Ophthalmic Solution 0.5% BID
Number analyzed (Participants) | 34 | 36 | 23
days | 224.4 (137.28) | 101.8 (105.69) | 314.6 (111.30)

ADVERSE EVENTS:
Time Frame: 1 year (12 months)
Arm/Group | AR-13324 Ophthalmic Solution 0.02% & Placebo | AR-13324 Ophthalmic Solution 0.02% BID | Timolol Maleate Ophthalmic Solution 0.5% BID
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/36 | 1/23
Other Adverse Events (participants affected / at risk) | 33/34 | 36/36 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=34) | AR-13324 Ophthalmic Solution 0.02% BID (N=36) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=23)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anterior Uveitis (Eye disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.02% & Placebo (N=34) | AR-13324 Ophthalmic Solution 0.02% BID (N=36) | Timolol Maleate Ophthalmic Solution 0.5% BID (N=23)
Conjunctival Hyperaemia (Eye disorders) | 28 | 34 | 2
Corneal Verticillata (Eye disorders) | 13 | 14 | 0
Erythema of Eyelid (Eye disorders) | 5 | 10 | 2
Conjunctival Haemorrhage (Eye disorders) | 7 | 6 | 0
Eyelid Oedema (Eye disorders) | 4 | 7 | 0
Lacrimation Increased (Eye disorders) | 7 | 4 | 0
Corneal Opacity (Eye disorders) | 5 | 4 | 0
Blepharitis (Eye disorders) | 2 | 5 | 0
Vision Blurred (Eye disorders) | 2 | 5 | 0
Conjunctival Oedema (Eye disorders) | 3 | 3 | 0
Eye Pruritis (Eye disorders) | 3 | 3 | 0
Eye Pain (Eye disorders) | 2 | 3 | 1
Eye Irritation (Eye disorders) | 1 | 3 | 0
Eyelids Pruritus (Eye disorders) | 1 | 3 | 0
Foreign Body Sensation in Eye (Eye disorders) | 0 | 4 | 0
Lenticular Opacities (Eye disorders) | 3 | 1 | 0
Conjunctivochalasis (Eye disorders) | 2 | 1 | 0
Eye Discharge (Eye disorders) | 2 | 1 | 0
Photophobia (Eye disorders) | 2 | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 2 | 0
Eye Allergy (Eye disorders) | 2 | 0 | 0
Eyelid Pain (Eye disorders) | 0 | 2 | 0
Optic Disc Haemorrhage (Eye disorders) | 0 | 2 | 1
Dry Eye (Eye disorders) | 1 | 0 | 2
Instillation Site Pain (General disorders) | 9 | 8 | 6
Instillation Site Discomfort (General disorders) | 6 | 2 | 1
Instillation Site Erythema (General disorders) | 2 | 2 | 0
Instillation Site Pruritus (General disorders) | 2 | 0 | 0
Vital Dye Staining Cornea Present (Investigations) | 14 | 8 | 7
Intraocular Pressure Increased (Investigations) | 3 | 1 | 0
Blood Triglycerides Increased (Investigations) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment was discontinued after 93 participants were enrolled due to slow enrollment; all participants who entered the study were followed until study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No